CLINICAL TRIAL: NCT01288755
Title: A Phase I, Open-label, Randomized, Crossover Trial in Healthy Subjects to Investigate the Pharmacokinetic Interaction Between TMC278 25 mg q.d. and Raltegravir 400 mg b.i.d.
Brief Title: TMC278-TiDP6-C153 - A Study in Healthy Volunteers Investigating the Pharmacokinetic Interaction Between TMC278 and Raltegravir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Collaborators: Raltegravir is provided by Merck. (Unknown)
Responsible Party: Compound Development Team Leader, Tibotec Pharmaceuticals, Ireland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR017773; TMC278-TiDP6-C153
Record Dates: First submitted 2011-01-07; First posted 2011-02-02 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: HIV Infections
Keywords: TMC278-TiDP6-C153; TMC278-C153; TMC278; HIV
MeSH Terms: conditions — HIV Infections | interventions — Rilpivirine; Raltegravir Potassium

ARMS (2):
- 001 (Experimental): TMC278 One 25 mg tablet once daily for 11 days (TrtA and C)
  Interventions: Drug: TMC278
- 002 (Experimental): Raltegravir One 400 mg tablet twice daily for 4 days (Trt B) and for 11 days (TrtC)
  Interventions: Drug: Raltegravir

INTERVENTIONS:
Drug: TMC278 — One 25 mg tablet, once daily, for 11 days (TrtA and C)
  Arms: 001
Drug: Raltegravir — One 400 mg tablet, twice daily, for 4 days (Trt B) and for 11 days (TrtC)
  Arms: 002

SUMMARY:
The purpose of this study is to investigate the effect of steady-state concentrations of raltegravir (administered as 400 mg, twice daily) on the steady-state pharmacokinetics of TMC278 (25 mg, once daily), and vice versa. Steady state is a term that means that the drug has been given long enough so that the plasma levels will remain at about the same level with each subsequent dose. TMC278 is being investigated for the treatment of human immunodeficiency virus (HIV) infection. Raltegravir is a commercially available antiretroviral drug for treatment of HIV infection. Pharmacokinetics (PK) means how the drug is absorbed into the bloodstream, distributed in the body and eliminated from the body.

DETAILED DESCRIPTION:
TMC278 is being investigated for treatment of HIV infection. Raltegravir is a commercially available HIV drug. The results of this study will provide dosing recommendations for coadministration of TMC278 and raltegravir in HIV-infected patients. This is a Phase I, open-label (both participant and investigator know the name of the medication given at a certain moment), randomized (sequence of treatment with study medications is assigned by chance), crossover trial in 24 healthy volunteers to investigate the pharmacokinetic interaction between TMC278 and raltegravir, at steady state. The study will consist of 3 phases: a screening phase, an open-label treatment phase consisting of 2 treatment periods, and end-of-study or withdrawal assessments. The duration of participation in the study for an individual participant will be up to 3 months (including screening). All participants will be randomly assigned to 1 of 2 possible treatment sequences and receive the following 2 treatments (Trt-s): TMC278 25 mg, once daily, alone for 11 days (TrtA), and raltegravir 400 mg, twice daily, alone for 4 days immediately followed by coadministration of the same raltegravir dose plus TMC278 25 mg, once daily, for 11 days (TrtB+C). There will be a washout period (a period where no study drug will be taken in view of having all the medication eliminated from the body before starting a new treatment) of at least 14 days between last intake of study medication in one session and first intake of study medication in the subsequent session. Pharmacokinetic profiles of both compounds will be determined through blood samples taken at regular intervals during the study. Safety and tolerability will be assessed during the study period and in follow-up. Blood and urine samples, electrocardiogram (ECG) and vital signs (blood pressure and heart rate) will be taken at screening, before medication intake in TrtA on Days 1, 11, and 12 (Day 12 is without ECG), in TrtB+C on Days 1, 4, 5, 15, and 16 (Day 16 is without ECG) and at the 2 follow-up visits (but without ECG) at 1 week and 4 weeks after last dose of study medication in the last session. A physical examination will be performed at screening, on Days 10 and 12 of TrtA, on Days 3, 14, and 16 of TrtB+C, and at both follow-up visits. Healthy volunteers will stay overnight in the study center for 3 nights in TrtA and for 5 nights in TrtB+C. Each volunteer will receive in a randomized order 2 treatments, minimum 14 days apart from each other. TrtA is TMC278 25 mg, once daily, for 11 days. TrtB+C is raltegravir 400 mg, twice daily, alone for first 4 days (TrtB) followed by coadministration of 400 mg raltegravir, twice daily, and TMC278 25 mg, once daily, on Days 5 to 15 (TrtC).

ELIGIBILITY:
Inclusion Criteria:

* Healthy, based on physical examination, medical history, vital signs, ECG, blood biochemistry, hematology and urinalysis
* Body Mass Index of 18 to 30.0 kg/m2
* Non-smoking for at least 3 months prior to screening
* Women must be postmenopausal for at least 2 years, or be surgically sterile.

Exclusion Criteria:

* Infected with Hepatitis A, B, or C Virus
* Infected with human immunodeficiency virus (HIV)
* History of clinically relevant hearth rhythm disturbances
* Having previously participated in more than 1 study with raltegravir, TMC125, TMC120 and/or TMC278 or having developed rash, erythema or urticaria while participating in a trial with aforementioned compounds

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-02; Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Change in exposure to TMC278 following co-administration with raltegravir and vice versa | Measured on Days 5, 12, 13, 14, 15, and 16 (TrtC). Reference for exposure to raltegravir only (TrtB), measured on Days 1, 2, 3, and 4. Reference for exposure to TMC278 only (TrtA), measured on Days 1, 8, 9, 10, 11, and 12.

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability - TMC278 and raltegravir. | 97 to 99 days (until and including last safety follow-up visit)

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited